CLINICAL TRIAL: NCT03184766
Title: An Open-label, Randomised, Three-way Cross-over, Single Dose, Single Centre, Comparative Pharmacokinetic Study Between Ibuprofen and Pseudoephedrine Liquid Capsules (2x 200 mg Ibuprofen & 30 mg Pseudoephedrine) (Test), Ibuprofen and Pseudoephedrine Tablets (2x 200 mg Ibuprofen & 30 mg Pseudoephedrine) (Comparator 1), and Ibuprofen Liquid Capsules (2x 200 mg Solubilised Ibuprofen) (Comparator 2)
Brief Title: Ibuprofen and Pseudoephedrine Comparative Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NL1309
Record Dates: First submitted 2017-05-17; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — Influenza Vaccines; Ibuprofen; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): Treatment Order: Test, Comparator 1, Comparator 2
  Interventions: Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules; Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets; Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules
- 2 (Experimental): Treatment Order: Test, Comparator 2, Comparator 1
  Interventions: Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules; Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets; Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules
- 3 (Experimental): Treatment Order: Comparator 1, Test, Comparator 2
  Interventions: Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules; Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets; Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules
- 4 (Experimental): Treatment Order: Comparator 1, Comparator 2, Test
  Interventions: Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules; Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets; Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules
- 5 (Experimental): Treatment Order: Comparator 2, Test, Comparator 1
  Interventions: Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules; Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets; Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules
- 6 (Experimental): Treatment Order: Comparator 2, Comparator 1, Test
  Interventions: Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules; Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets; Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules

INTERVENTIONS:
Drug: Test Nurofen Cold and Flu®, Ibuprofen and pseudoephedrine liquid capsules — 2 x 200 mg ibuprofen & 30 mg pseudoephedrine
Drug: Comparator 1 Nurofen Cold and Flu®, ibuprofen and pseudoephedrine tablets — 2 x 200 mg ibuprofen & 30 mg pseudoephedrine
Drug: Comparator 2 Nurofen Immedia 200 mg Weichkapseln, ibuprofen liquid capsules — 2 x 200 mg solubilised ibuprofen

SUMMARY:
This comparative pharmacokinetic study is being conducted to provide supporting evidence for inclusion in dossiers to regulatory authorities for an Article 8(3) of Directive 2001/83/EC abridged application for ibuprofen and pseudoephedrine liquid capsules (200 mg ibuprofen & 30 mg pseudoephedrine).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who have given written informed consent.
2. Age: ≥ 18 years ≤ 50 years.
3. Body Mass Index (BMI) of ≥ 20 and ≤ 30 kg/m2.
4. Healthy as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
5. Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use an effective method of contraception unless of non-childbearing potential or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject from first dose until 3 months after the final dose of study medication.
6. Female subject of non-child bearing potential with negative pregnancy test at the screening visit.
7. Male subject willing to use an effective method of contraception unless anatomically sterile or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject from first dose until 3 months after the final dose of study medication.

Exclusion Criteria:

1. Pregnant or lactating females.
2. A history and/or presence of significant disease of any body system, including psychiatric disorders.
3. Any condition that may currently interfere with the absorption, distribution, metabolism or excretion of drugs.
4. A history of allergy or intolerance related to treatment with ibuprofen, aspirin, other NSAIDs, pseudoephedrine, other sympathomimetic or catecholamine derivative decongestant drugs or the excipients of the formulations.
5. A history of or active peptic or duodenal ulcers or gastro-intestinal bleed or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders.
6. A history of hypertension or hypertension that is currently treated with antihypertensive medication.
7. A history of frequent dyspepsia, e.g. heartburn or indigestion.
8. A history of migraine.
9. Current smokers and ex-smokers who have smoked or used nicotine replacement products during the previous 6 months prior to first dosing.
10. A history of substance abuse (including alcohol).
11. High consumption of stimulating drinks (coffee, tea, cola, energy drinks etc.; total caffeine intake per day above 300 mg).
12. Those with positive screen/test for drugs of abuse and alcohol.
13. Those with a positive screen for ibuprofen.
14. Ingestion of a prescribed drug at any time in the 14 days before the first dose of study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers 30 days prior to the first dose of study medication.
15. Ingestion of an over-the-counter preparation within 7 days before the first dose of study medication, including herbal medications, vitamin/fish oil supplements, ibuprofen, other NSAIDs or decongestants.
16. Donation of blood in quantity > 400 ml e.g. to the blood transfusion service in the 12 weeks prior to the first dose of study medication
17. Known human immune deficiency virus (HIV) positive status, or a positive viral serology screen.
18. Topical use of ibuprofen within 7 days before the first dose of study medication.
19. Those previously randomised into this study.
20. Those who are an employee at the study site.
21. Those who are a partner or first degree relative of the Investigator.
22. Those who have participated in a clinical trial in the 12 weeks prior to the first dose of study medication.
23. Those unable in the opinion of the Investigator to comply fully with the study requirements.
24. Those who have consumed grapefruit or grapefruit juice, pummelo or Seville oranges in the 7 days prior to randomisation.
25. Those who are unwilling to consume gelatine of animal origin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Pseudoephedrine AUC0-t for Test vs. Comparator 1. | PK Analysis: 0-48hrs
  The Test and Comparator 1 will be considered similar if for pseudoephedrine, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator 1 ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Pseudoephedrine Cmax for Test vs. Comparator 1. | PK Analysis: 0-48hrs
  The Test and Comparator 2 will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator 2 ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Ibuprofen AUC0-t for Test vs. Comparator 2. | PK Analysis: 0-48hrs
  The Test and Comparator 2 will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator 2 ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Ibuprofen Cmax for Test vs. Comparator 2. | PK Analysis: 0-48hrs
  The Test and Comparator 2 will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator 2 ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:

SECONDARY OUTCOMES:
Ibuprofen AUC0-t for Test vs. Comparator 1. | PK Analysis: 0-48hrs
  The Test and Comparator 1 will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator 1 ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
  • Cmax for ibuprofen (in the context of the Test vs. Comparator 1 comparison)
Ibuprofen Cmax for Test vs. Comparator 1. | PK Analysis: 0-48hrs
  The Test and Comparator 1 will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator 1 ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Assessment of how fast the ibuprofen from the Test product starts to be absorbed and how quickly it reaches the therapeutic level. | PK Analysis: 0-48hrs
  T8.4 - time to reach the therapeutic level (8.4 µg/ml) for ibuprofen.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  Cn - the plasma concentration of an active at each planned nominal time-point.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  AUC0-inf - Area under the plasma concentration-time curve from administration to infinity.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  administration to infinity. AUCR - ratio AUC0-t / AUC0-inf.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  Tmax -Time until Cmax is first achieved.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  Kel - elimination rate constant.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  T1/2 - plasma concentration half-life.
Pharmacokinetic parameters will be assessed as secondary endpoints. | PK Analysis: 0-48hrs
  Tlag - time between administration and the beginning of absorption of ibuprofen. This will be calculated only for the Test.

OTHER OUTCOMES:
The occurrence of Adverse Events. | Through study completion - Screening to study follow-up (Approx 8 weeks)
Change from baseline in oral temperature. | Through study completion - Screening to study follow-up (Approx 8 weeks)
  Measured in degrees Celcius
Change from baseline in resting heart rate. | Through study completion - Screening to study follow-up (Approx 8 weeks)
  Measured in beats per minute
Change from baseline in resting blood pressure. | Through study completion - Screening to study follow-up (Approx 8 weeks)
  Measured in mmHg
Change from baseline in haematology testing. | Through study completion - Screening to study follow-up (Approx 8 weeks)
Change from baseline in biochemistry testing. | Through study completion - Screening to study follow-up (Approx 8 weeks)
Change from baseline in urinary testing. | Through study completion - Screening to study follow-up (Approx 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Adams, MBBS, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: No